CLINICAL TRIAL: NCT06544252
Title: Pre-exercise Ingestion of a Low Glycaemic Index Rice-based Mixed Meal Increases Fat Oxidation and Endurance Running in a Hot-humid Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Zaini Bahari, Principle Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/19010083
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Trained Athletes

STUDY DESIGN:
Intervention Model Description: The present study employed a randomised, single-blind, cross-over trial design consisting of two experimental trials separated by a one-week washout period to minimise carryover effects, conducted under hot-humid (32°C, 65% RH) conditions.. The participants were randomised into two groups, each comprising six participants. Six participants were randomised to receive low glycaemic index, and the other six participants received high glycaemic index pre-exercise dietary interventions, followed by a cross-over with the opposing dietary intervention after one week.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low glycaemic index, Then high glycaemic index (Experimental): The participants were randomised to receive pre-exercise low glycaemic index rice-based mixed meal followed by a cross-over with the high glycaemic index rice-based mixed meal after one week
  Interventions: Dietary Supplement: Low glycaemic index rice-based mixed meal (GI value = 47); Dietary Supplement: High glycaemic index rice-based mixed meal (GI value = 80)
- High glycaemic index, Then low glycaemic index (Experimental): The participants were randomised to receive pre-exercise high glycaemic index rice-based mixed meal followed by a cross-over with the low glycaemic index rice-based mixed meal after one week
  Interventions: Dietary Supplement: Low glycaemic index rice-based mixed meal (GI value = 47); Dietary Supplement: High glycaemic index rice-based mixed meal (GI value = 80)

INTERVENTIONS:
Dietary Supplement: Low glycaemic index rice-based mixed meal (GI value = 47) — The mixed meal consisted of Basmati rice, chicken, and green-leafy vegetables. The energy content of the mixed meal was based on the body mass of the participant. The amount of CHO was 1.3 g.kg-1 body mass (Burke et al. 2019), and the amount of protein given was 0.5 g.kg-1 per meal (Witard, Garthe and Phillips 2019).
Dietary Supplement: High glycaemic index rice-based mixed meal (GI value = 80) — The mixed meal consisted of fragrant rice, chicken, and green-leafy vegetables.The energy content of the mixed meal was based on the body mass of the participant. The amount of CHO was 1.3 g.kg-1 body mass (Burke et al. 2019), and the amount of protein given was 0.5 g.kg-1 per meal (Witard, Garthe and Phillips 2019).

SUMMARY:
The objective of this research is to determine the influence of low and high glycemic index Malaysian pre-exercise mixed meals on endurance exercise performance in a hot-humid environment. Glycemic index (GI) is a method used to classify CHO-containing foods based on their influence on postprandial blood glucose when compared to the response on blood glucose after ingesting the same amount of CHO from a reference food (glucose or bread). Low GI (LGI) foods are digested and absorbed more slowly as compared to high GI (HGI) foods, resulting in a stable rise in blood glucose levels.

The participants were trained male endurance long-distance runners. On the day of experimental trials, they consumed pre-exercise rice-based mixed meal, either LGI or HGI 3 hours before endurance running exercise. After that, they ran for 45 minutes at constant running speed equivalent to 70% VO2peak, followed by 10km time-trial. The respiratory gases, blood measures, rectal and skin temperature were measured throughout the running test.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 18-35 years old
* trained (peak oxygen consumption (V̇O2peak): ≥ 55 mL.kg-1.min-1)
* training volume (>150 min, ≥ three times per week)
* competing at the national level
* >2-year of running experience
* tier 2 (trained) or tier 3 (highly trained) runners (McKay et al. 2022)
* no allergies to any test foods

Exclusion Criteria:

* diagnosis of chronic diseases (i.e. diabetes mellitus, hypertension, cardiovascular disease)
* bone, muscle or joint impairments
* on medication
* currently smoking
* use of illicit drugs
* use of dietary supplements
* on any particular diet

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Time to complete 10 km time-trial | Up to 1 hour
  The participant was clearly instructed to complete the 10 km time-trial as quickly as possible. The 10 km time-trial commenced with a 30-s rolling start to the participant's 70% V̇O2peak speed, after which the participant could freely adjust the speed. Throughout the 10 km time-trial, the prevailing running velocity and time-lapse were blinded to the participant, and only information on the distance covered at 1 km intervals was verbally provided to the participant.

SECONDARY OUTCOMES:
Fat and carbohydrate oxidation | Up to 2 hours
  A portable gas analyser (K5, COSMED, Italy) was used to measure the respiratory gas exchange. Prior to each experimental session, the device was calibrated according to the procedures outlined in the manufacturer's instructions. The mixing chamber measurements were performed for V̇O2, V̇CO2, and respiratory exchange ratio (RER) and were measured continuously throughout exercise trials. The average values for V̇O2 (L.min-1) and V̇CO2 (L.min-1) were calculated over the last 30-s of each 15-min interval during SS running and each 1 km of 10 km time-trial.
  Whole-body rates of CHO and fat oxidation (g.min-1) were calculated using intensity-dependent equations for moderate to high-intensity exercise (50 - 75% V̇O2max) that assume negligible protein contribution to energy expenditure (Jeukendrup and Wallis 2005):
  CHO oxidation (g.min-1): (4.210 x V̇CO2) - (2.962 x V̇O2) Fat oxidation (g.min-1): (1.695 x V̇O2) - (1.701 x V̇CO2)
Capillary blood glucose | Up to 5 hours
  The capillary blood was sampled for blood glucose via a finger prick using a sterile, single-use lancet (Accu-Check Safe-T-Pro Plus; Roche Diagnostics) during fasting state (before meal consumption), postprandial period (at 15, 30, 60, 90, 120, 180-min intervals), steady-state running (at 10, 30, 45-min intervals), time-trial 10km running performance (at 5, 10km marks).
Serum insulin | Up to 5 hours
  The venous blood was sampled for insulin using 22G IV catheter insertion (Surflo IV Catheter, Terumo Med Corporation, Eklton, MD., USA) during fasting state (before meal consumption), postprandial period (at 30, 90, 180-min intervals), steady-state running (at 10, 30, 45-min intervals), time-trial 10km running performance (at 10 km marks).
Serum cortisol | Up to 5 hours
  The venous blood was sampled for cortisol using 22G IV catheter insertion (Surflo IV Catheter, Terumo Med Corporation, Eklton, MD., USA) during fasting state (before meal consumption), postprandial period (at 180-min interval), steady-state running (at 45-min interval), time-trial 10km running performance (at 10 km marks).
Serum lactate | Up to 2 hours
  The venous blood was sampled for lactate using 22G IV catheter insertion (Surflo IV Catheter, Terumo Med Corporation, Eklton, MD., USA) at postprandial period (at 180-min interval), steady-state running (at 10, 45-min intervals), time-trial 10 km running performance (at 10 km marks).
Heart rate | Up to 2 hours
  Heart rate was recorded using heart rate monitor (Garmin HRM-Run®; Olathe, KS, USA) throughout the running test.
Thermoregulatory measure | Up to 2 hours
  Rectal temperature (Tre), and skin temperature (Tsk) were continuously measured throughout the running exercise. Tre was measured by self-inserting a disposable thermistor probe (YSI 400 series, Mallinckrodt Medical, Kansas City, Mo., USA) 12 cm beyond the anal sphincter. Tsk was assessed at four distinct sites (left shoulder, left chest, right mid-thigh, and right mid-shin) using iButton temperature sensors (Maxim Integrated Products,Sunnyvale, CA., USA).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Munir Che Muhamed, PhD, Principal Investigator — Department of Community Health, Advanced Medical and Dental Institute, Universiti Sains Malaysia, Bertam, 13200, Kepala Batas, Pulau Pinang, Malaysia
Locations (1):
- Department of Community Health, Advanced Medical and Dental Institute, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Private and confidential